CLINICAL TRIAL: NCT04363775
Title: Comparison of VieScope Versus Macintosh Laryngoscope for Emergency Intubation Under Level C Personal Protective Equipment Conditions
Brief Title: Comparison of VieScope vs. Macintosh Laryngoscope for Intubation in Level Cpersonal Protective Equipment Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Collaborators: Poznan University of Medical Sciences (Other); Wroclaw Medical University (Other); Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Associate Profesor, Lazarski University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: INT_PPE_2020_1
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Tracheal Intubation; Infection; Projection
Keywords: SARS-CoV-2; COVID-19; tracheal intubation; laryngoscope; personal protective equipment
MeSH Terms: conditions — Infections; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regurgitation (Experimental): intubation in regurgitation condition
  Interventions: Device: The standard Macintosh laryngoscope; Device: The Vie Scope laryngoscope
- Tongue edema (Experimental): intubation in Tongue edema condition
  Interventions: Device: The standard Macintosh laryngoscope; Device: The Vie Scope laryngoscope

INTERVENTIONS:
Device: The standard Macintosh laryngoscope — intubation with the standard Macintosh laryngoscope and endotracheal tube 7.0 internal diameter with standard tube stylet
  Other Names: MAC
Device: The Vie Scope laryngoscope — intubation with the Vie Scope laryngoscope with bougie stylet and endotracheal tube 7.0 internal diameter
  Other Names: VSCOPE

SUMMARY:
The current COVID-19 pandemic, this is especially since the transmission of SARS-CoV-2 is thought to occur mainly through respiratory droplets generated by coughing and sneezing, by direct contact with contaminated surfaces and because in a large number of patients COVID-19 disease may be asymptomatic. As recommended by the CDC for aerosol-generating procedures (AGP), medical personnel should be equipped with full personal protective equipment (PPE) for AGP. Therefore, it is reasonable to search for the most effective methods of intubation in those conditions.

ELIGIBILITY:
Inclusion Criteria:

* paramedic
* consent voluntary participation in the study
* none experience in Vie Scope
* none experience in intubation with personal protective equipment

Exclusion Criteria:

* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-02-23 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
time to intubation | 1 day
  time from pick up device to the final placement tube in trachea

SECONDARY OUTCOMES:
success of intubation | 1 day
  A failed intubation attempt was defined as an attempt in which the trachea was not intubated, or which required more than 120 seconds to perform
Number of optimalization maneuvers | 1 day
  the number of optimization maneuvers required (re-adjustment of head position, second assistant) to aid endotracheal intubation
Procedure Ease of use | 1 day
  self-reported percentage the vocal cord visualization. A 100% score is a extremely difficult procedure. A Ease of use score of 1% means that procedure is extremely easy
the degree of visibility of the glottis | 1 day
  The POGO score describes how much glottic opening is visible. A POGO score of 100% indicates visualization of the entire glottic opening from the anterior commissure of the vocal cords to the interarytenoid notch. A POGO score of 0% corresponds with no visualization of laryngeal structures.
Cormack - Lehane grade | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)

CONTACTS AND LOCATIONS:
Locations (1):
- Lazarski Univeristy, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
we will decided after finishing manuscript